CLINICAL TRIAL: NCT04605406
Title: Daily Step Count and Achieving Goal Gestational Weight Gain
Status: Withdrawn | Type: Observational
Why Stopped: No participants recruited for the study.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Serdar Ural, Associate Professor of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Other Study IDs: STUDY00014096
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related
Keywords: pregnant; pregnancy; gestational weight; weight gain; gestational weight gain
MeSH Terms: conditions — Weight Gain; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this voluntary research study is to determine an optimal step count that aids in achieving the recommended weight gain during pregnancy and to use this count in future studies.

DETAILED DESCRIPTION:
The goal of this study is to contribute to the growing data that show a clear benefit in activity during pregnancy over sedentary behavior. Uniquely, this study looks to determine an optimal step count for achieving goal gestational weight gain. In doing so, this will enable clinicians to better counsel patients on a low cost, at home activity that can aid in improved maternal and fetal outcomes. This optimal step count would be used in future randomized clinical trials to determine whether this goal step count could be used to benefit other maternal and fetal outcomes such as gestational diabetes, preeclampsia, preterm labor, cesarean section rates, and birth weight.

Participation will begin at the patients 18-22 week clinic visit and will last until delivery. At the 18 - 22 week clinic visit a pedometer will be given to the patient. Patient will be instructed by a study team member to wear the pedometer on a hip for 7 days every 4 weeks and will submit daily step count for the day via a link to an online submission form which will arrive in the email once a day for 7 days in a row. An email reminder will be received every four weeks to prepare the patient for the reporting of daily step count, if no response is received electronically via the online submission form after 14 days a second reminder will be received. No change in normal activity will be required, instructions will be given to maintain normally activity during the week. The pedometer will be returned when patient arrives to labor and delivery to deliver.

The risks of this study are minimal as there will be no diversion from normal daily routine.

The results of this research may guide the future studies in walking in pregnancy in relation to maternal, fetal, and neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Pregnant women
3. A singleton pregnancy
4. Gestational age at inclusion 18-22 weeks
5. Ability to read and speak English
6. Access to a computer
7. Cell phone

Exclusion Criteria:

1. Multiple pregnancy
2. Pregestational diabetes
3. Diseases limiting level of physical activity
4. Previous bariatric surgery
5. Current alcohol use
6. Current drug abuse
7. Currently in a opioid treatment program
8. History of eating disorder
9. Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Recruited at the time of their 18-22 week second trimester ultrasound in the Obstetrics and Gynecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimal average steps per day to achieve goal GWG | Steps per day will be measured for 7 consecutive days every 4 weeks after enrollment at the 18-22 week clinic visit until delivery at 37-41 weeks.
  Assessing the optimal average steps per day a pregnant woman should take to meet her goal gestational weight gain (GWG) based on ACOG guidelines. Meeting the goal GWG is defined as a yes/no response.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Ural, MD, Principal Investigator — Penn State Health
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of IPD will only be permitted when contact has been made with the Principal Investigator, Dr. Serdar Ural, and once request access to the dataset has been approved.
Supporting Information: Study Protocol
Time Frame: Length of time to complete the outcomes, estimating 6 months.

REFERENCES:
- [Background] Kominiarek MA, Balmert LC, Tolo H, Grobman W, Simon M. A feasibility study of activity tracking devices in pregnancy. BMC Pregnancy Childbirth. 2019 Nov 4;19(1):401. doi: 10.1186/s12884-019-2557-3. PMID 31684889
- [Background] Kong KL, Campbell CG, Foster RC, Peterson AD, Lanningham-Foster L. A pilot walking program promotes moderate-intensity physical activity during pregnancy. Med Sci Sports Exerc. 2014 Mar;46(3):462-71. doi: 10.1249/MSS.0000000000000141. PMID 24002348
- [Background] Ferrari RM, Siega-Riz AM, Evenson KR, Moos MK, Carrier KS. A qualitative study of women's perceptions of provider advice about diet and physical activity during pregnancy. Patient Educ Couns. 2013 Jun;91(3):372-7. doi: 10.1016/j.pec.2013.01.011. Epub 2013 Feb 9. PMID 23399436
- [Background] Connolly CP, Coe DP, Kendrick JM, Bassett DR Jr, Thompson DL. Accuracy of physical activity monitors in pregnant women. Med Sci Sports Exerc. 2011 Jun;43(6):1100-5. doi: 10.1249/MSS.0b013e3182058883. PMID 21085037
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee opinion no. 548: weight gain during pregnancy. Obstet Gynecol. 2013 Jan;121(1):210-2. doi: 10.1097/01.aog.0000425668.87506.4c. PMID 23262962
- [Background] Kominiarek MA, Vyhmeister H, Balmert LC, Fairchild P, Tolo H, Grobman W, Simon M. Activity Tracking Devices in Group Prenatal Care: A Feasibility Study. Biores Open Access. 2018 Nov 28;7(1):165-176. doi: 10.1089/biores.2018.0021. eCollection 2018. PMID 30505631
- [Background] Kinnunen TI, Tennant PW, McParlin C, Poston L, Robson SC, Bell R. Agreement between pedometer and accelerometer in measuring physical activity in overweight and obese pregnant women. BMC Public Health. 2011 Jun 27;11:501. doi: 10.1186/1471-2458-11-501. PMID 21703033
- [Background] Cohen TR, Plourde H, Koski KG. Are Canadian women achieving a fit pregnancy? A pilot study. Can J Public Health. 2010 Jan-Feb;101(1):87-91. doi: 10.1007/BF03405570. PMID 20364546
- [Background] Skreden M, Overby NC, Sagedal LR, Vistad I, Torstveit MK, Lohne-Seiler H, Bere E. Change in active transportation and weight gain in pregnancy. Int J Behav Nutr Phys Act. 2016 Jan 27;13:10. doi: 10.1186/s12966-016-0332-7. PMID 26818593
- [Background] Westgarth C, Liu J, Heron J, Ness AR, Bundred P, Gaskell RM, German AJ, McCune S, Dawson S. Dog ownership during pregnancy, maternal activity, and obesity: a cross-sectional study. PLoS One. 2012;7(2):e31315. doi: 10.1371/journal.pone.0031315. Epub 2012 Feb 15. PMID 22355356
- [Background] Cremona A, O'Gorman C, Cotter A, Saunders J, Donnelly A. Effect of exercise modality on markers of insulin sensitivity and blood glucose control in pregnancies complicated with gestational diabetes mellitus: a systematic review. Obes Sci Pract. 2018 Sep 4;4(5):455-467. doi: 10.1002/osp4.283. eCollection 2018 Oct. PMID 30338116
- [Background] McMillan AG, May LE, Gaines GG, Isler C, Kuehn D. Effects of Aerobic Exercise during Pregnancy on 1-Month Infant Neuromotor Skills. Med Sci Sports Exerc. 2019 Aug;51(8):1671-1676. doi: 10.1249/MSS.0000000000001958. PMID 30817721
- [Background] Lemmens PMC, Sartor F, Cox LGE, den Boer SV, Westerink JHDM. Evaluation of an activity monitor for use in pregnancy to help reduce excessive gestational weight gain. BMC Pregnancy Childbirth. 2018 Jul 31;18(1):312. doi: 10.1186/s12884-018-1941-8. PMID 30064390
- [Background] Bo K, Artal R, Barakat R, Brown W, Davies GA, Dooley M, Evenson KR, Haakstad LA, Henriksson-Larsen K, Kayser B, Kinnunen TI, Mottola MF, Nygaard I, van Poppel M, Stuge B, Khan KM. Exercise and pregnancy in recreational and elite athletes: 2016 evidence summary from the IOC expert group meeting, Lausanne. Part 1-exercise in women planning pregnancy and those who are pregnant. Br J Sports Med. 2016 May;50(10):571-89. doi: 10.1136/bjsports-2016-096218. No abstract available. PMID 27127296
- [Background] Bo K, Artal R, Barakat R, Brown W, Dooley M, Evenson KR, Haakstad LAH, Larsen K, Kayser B, Kinnunen TI, Mottola MF, Nygaard I, van Poppel M, Stuge B, Davies GAL; IOC Medical Commission. Exercise and pregnancy in recreational and elite athletes: 2016 evidence summary from the IOC expert group meeting, Lausanne. Part 2-the effect of exercise on the fetus, labour and birth. Br J Sports Med. 2016 Nov;50(21):1297-1305. doi: 10.1136/bjsports-2016-096810. Epub 2016 Oct 12. PMID 27733352
- [Background] Berghella V, Saccone G. Exercise in pregnancy! Am J Obstet Gynecol. 2017 Apr;216(4):335-337. doi: 10.1016/j.ajog.2017.01.023. Epub 2017 Feb 22. No abstract available. PMID 28236414
- [Background] Shieh C, Yang Z, Haas DM, Carpenter JS. Feasibility and Potential Benefits of a Self-Monitoring Enhanced Lifestyle Intervention to Prevent Excessive Gestational Weight Gain in Women Who Are Overweight or Obese. J Obstet Gynecol Neonatal Nurs. 2017 Mar-Apr;46(2):182-196. doi: 10.1016/j.jogn.2016.09.006. Epub 2017 Jan 5. PMID 28063804
- [Background] Chandonnet N, Saey D, Almeras N, Marc I. French Pregnancy Physical Activity Questionnaire compared with an accelerometer cut point to classify physical activity among pregnant obese women. PLoS One. 2012;7(6):e38818. doi: 10.1371/journal.pone.0038818. Epub 2012 Jun 11. PMID 22701717
- [Background] Kominiarek MA, Peaceman AM. Gestational weight gain. Am J Obstet Gynecol. 2017 Dec;217(6):642-651. doi: 10.1016/j.ajog.2017.05.040. Epub 2017 May 24. PMID 28549978
- [Background] Kong KL, Campbell C, Wagner K, Peterson A, Lanningham-Foster L. Impact of a walking intervention during pregnancy on post-partum weight retention and infant anthropometric outcomes. J Dev Orig Health Dis. 2014 Jun;5(3):259-67. doi: 10.1017/S2040174414000117. PMID 24901666
- [Background] Cohen TR, Koski KG. Limiting excess weight gain in healthy pregnant women: importance of energy intakes, physical activity, and adherence to gestational weight gain guidelines. J Pregnancy. 2013;2013:787032. doi: 10.1155/2013/787032. Epub 2013 Feb 20. PMID 23533762
- [Background] Harrison CL, Thompson RG, Teede HJ, Lombard CB. Measuring physical activity during pregnancy. Int J Behav Nutr Phys Act. 2011 Mar 21;8:19. doi: 10.1186/1479-5868-8-19. PMID 21418609
- [Background] Haby K, Berg M, Gyllensten H, Hanas R, Premberg A. Mighty Mums - a lifestyle intervention at primary care level reduces gestational weight gain in women with obesity. BMC Obes. 2018 Jun 4;5:16. doi: 10.1186/s40608-018-0194-4. eCollection 2018. PMID 29881627
- [Background] Haby K, Glantz A, Hanas R, Premberg A. Mighty Mums - An antenatal health care intervention can reduce gestational weight gain in women with obesity. Midwifery. 2015 Jul;31(7):685-92. doi: 10.1016/j.midw.2015.03.014. Epub 2015 Apr 9. PMID 25912510
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras V, Gray C, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater L, Stirling D, Zehr L. No. 367-2019 Canadian Guideline for Physical Activity throughout Pregnancy. J Obstet Gynaecol Can. 2018 Nov;40(11):1528-1537. doi: 10.1016/j.jogc.2018.07.001. Epub 2018 Oct 5. PMID 30297272
- [Background] DiNallo JM, Downs DS, Le Masurier G. Objectively assessing treadmill walking during the second and third pregnancy trimesters. J Phys Act Health. 2012 Jan;9(1):21-8. doi: 10.1123/jpah.9.1.21. PMID 22232501
- [Background] McParlin C, Robson SC, Tennant PW, Besson H, Rankin J, Adamson AJ, Pearce MS, Bell R. Objectively measured physical activity during pregnancy: a study in obese and overweight women. BMC Pregnancy Childbirth. 2010 Nov 29;10:76. doi: 10.1186/1471-2393-10-76. PMID 21114834
- [Background] Renault K, Norgaard K, Secher NJ, Andreasen KR, Baldur-Felskov B, Nilas L. Physical activity during pregnancy in normal-weight and obese women: compliance using pedometer assessment. J Obstet Gynaecol. 2012 Jul;32(5):430-3. doi: 10.3109/01443615.2012.668580. PMID 22663312
- [Background] Renault K, Norgaard K, Andreasen KR, Secher NJ, Nilas L. Physical activity during pregnancy in obese and normal-weight women as assessed by pedometer. Acta Obstet Gynecol Scand. 2010 Jul;89(7):956-61. doi: 10.3109/00016341003792459. PMID 20583938
- [Background] Medek H, Halldorsson T, Gunnarsdottir I, Geirsson RT. Physical activity of relatively high intensity in mid-pregnancy predicts lower glucose tolerance levels. Acta Obstet Gynecol Scand. 2016 Sep;95(9):1055-62. doi: 10.1111/aogs.12931. Epub 2016 Jun 9. PMID 27228200
- [Background] Nascimento SL, Surita FG, Godoy AC, Kasawara KT, Morais SS. Physical Activity Patterns and Factors Related to Exercise during Pregnancy: A Cross Sectional Study. PLoS One. 2015 Jun 17;10(6):e0128953. doi: 10.1371/journal.pone.0128953. eCollection 2015. PMID 26083416
- [Background] Bacchi E, Bonin C, Zanolin ME, Zambotti F, Livornese D, Dona S, Tosi F, Baldisser G, Ihnatava T, Di Sarra D, Bonora E, Moghetti P. Physical Activity Patterns in Normal-Weight and Overweight/Obese Pregnant Women. PLoS One. 2016 Nov 9;11(11):e0166254. doi: 10.1371/journal.pone.0166254. eCollection 2016. PMID 27829017
- [Background] Materia FT, Smyth JM, Heron KE, Hillemeier M, Feinberg ME, Fonzi P, Symons Downs D. Preconceptional health behavior change in women with overweight and obesity: prototype for SMART strong healthy women intervention. Mhealth. 2018 Jul 6;4:24. doi: 10.21037/mhealth.2018.06.06. eCollection 2018. PMID 30148139
- [Background] Yeo S, Logan JG. Preventing obesity: exercise and daily activities of low-income pregnant women. J Perinat Neonatal Nurs. 2014 Jan-Mar;28(1):17-25. doi: 10.1097/JPN.0000000000000000. PMID 24476648
- [Background] Shieh C, Draucker CB. Self-monitoring Lifestyle Behavior in Overweight and Obese Pregnant Women: Qualitative Findings. Clin Nurse Spec. 2018 Mar/Apr;32(2):81-89. doi: 10.1097/NUR.0000000000000355. PMID 29419580
- [Background] Dodd JM, Cramp C, Sui Z, Yelland LN, Deussen AR, Grivell RM, Moran LJ, Crowther CA, Turnbull D, McPhee AJ, Wittert G, Owens JA, Robinson JS; LIMIT Randomised Trial Group. The effects of antenatal dietary and lifestyle advice for women who are overweight or obese on maternal diet and physical activity: the LIMIT randomised trial. BMC Med. 2014 Oct 13;12:161. doi: 10.1186/s12916-014-0161-y. PMID 25315237
- [Background] Baruth M, Schlaff RA, Deere S, Walker JL, Dressler BL, Wagner SF, Boggs A, Simon HA. The Feasibility and Efficacy of a Behavioral Intervention to Promote Appropriate Gestational Weight Gain. Matern Child Health J. 2019 Dec;23(12):1604-1612. doi: 10.1007/s10995-019-02812-6. PMID 31541375
- [Background] Renault KM, Norgaard K, Nilas L, Carlsen EM, Cortes D, Pryds O, Secher NJ. The Treatment of Obese Pregnant Women (TOP) study: a randomized controlled trial of the effect of physical activity intervention assessed by pedometer with or without dietary intervention in obese pregnant women. Am J Obstet Gynecol. 2014 Feb;210(2):134.e1-9. doi: 10.1016/j.ajog.2013.09.029. Epub 2013 Sep 20. PMID 24060449
- [Background] Cohen TR, Plourde H, Koski KG. Use of the Pregnancy Physical Activity Questionnaire (PPAQ) to identify behaviours associated with appropriate gestational weight gain during pregnancy. J Phys Act Health. 2013 Sep;10(7):1000-7. doi: 10.1123/jpah.10.7.1000. Epub 2012 Nov 5. PMID 23132834
- [Background] Viecceli C, Remonti LR, Hirakata VN, Mastella LS, Gnielka V, Oppermann ML, Silveiro SP, Reichelt AJ. Weight gain adequacy and pregnancy outcomes in gestational diabetes: a meta-analysis. Obes Rev. 2017 May;18(5):567-580. doi: 10.1111/obr.12521. Epub 2017 Mar 8. PMID 28273690